CLINICAL TRIAL: NCT03998917
Title: Pathophysiological Characterization of the Neuromuscular Function of a Population With Multiple Comorbidities Suffering From Chronic Renal Failure in Pre-dialysis.
Acronym: PIONNIER
Status: Withdrawn | Type: Observational
Why Stopped: Human subjects protection's soubmission denied
Sponsor: Centre Hospitalier le Mans (Other)
Collaborators: Le Mans Universite (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2019/S8/02
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Failure; Chronic Kidney Disease stage3; Chronic Kidney Disease, Stage 4 (Severe); Chronic Kidney Disease Stage 5; Fatigue
Keywords: Chronic Kidney Failure; Fatigue; Adapted Physical Activity
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease (CKD) Patients: Patients with chronic kidney disease and a glomerular filtration rate less than 60 ml/min of creatinine. Patients will perform a hand grip fatigability test with their dominant hand, followed by a Timed Up and Go Test (TUG-Test), a Five-repetition sit-to-stand-test (5STS-Test) and a10 meters gait speed test.
  Interventions: Diagnostic Test: Discrimination of neuromuscular alterations protocol
- Control cohort: The control cohort will consist of a group of people from the same age group as the CKD group but without chronic kidney disease. The exclusion criteria apply to this group. They will be selected from the spouses and other volunteers. This group will also perform a hand grip fatigability test with their dominant hand, followed by a Timed Up and Go Test (TUG-Test), a Five-repetition sit-to-stand-test (5STS-Test) and a10 meters gait speed test.
  Interventions: Diagnostic Test: Discrimination of neuromuscular alterations protocol

INTERVENTIONS:
Diagnostic Test: Discrimination of neuromuscular alterations protocol — Patients will perform a hand grip fatigability test with their dominant hand, followed by a Timed Up and Go Test (TUG-Test), a Five-repetition sit-to-stand-test (5STS-Test) and a10 meters gait speed test.

SUMMARY:
The evolution of chronic kidney disease (CKD) causes a systemic upheaval on the body and a deep fatigue is very often described by patients (50-70% of the patients) even before the start of dialysis (pre-dialysis). This fatigue has many origins, and one of them probably stems from a deterioration of neuromuscular abilities. Very few studies have examined the physiological aspects of neuromuscular fatigue in pre-dialysis patients, and shedding light on potential deficits at this level would allow safe and efficient implementation of adapted physical activity programs.

Our study aims to characterize the pathophysiology of neuromuscular capabilities in chronic advanced renal failure in pre-dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age> 18 years) who have signed the informed consent form
* Social security coverage
* For patients in the Chronic Kidney Disease group: Glomerular filtration rate less than 60 ml/min of creatinine for more than three months

Exclusion Criteria:

* Dermatological conditions of the upper limbs which would contra-indicate Electromyographic electrodes being positioned
* Gestating women
* Patients with known neuromuscular conditions
* Patients with dementia
* Patients with acute heart failure
* Patients with a history of surgery of the evaluated limb
* Patients included in an interventional study involving administration of treatments other than routine care
* For the patients in the Chronic Kidney Disease group: patients currently undergoing dialysis or in a pre-dialysis program (e.g. with a dialysis fistula already in place).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Kidney Disease (CKD) group:
  Patients with chronic kidney disease and a glomerular filtration rate less than 60 ml/min of creatinine.
  Control group:
  The control group will consist of a group of people from the same age group as the CKD group but without chronic kidney disease. The exclusion criteria apply to this group. They will be selected from the spouses and other volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular evaluation of force. | 1 day
  Maximum force normalized by body mass, measured by a hand grip test with the dominant hand.

SECONDARY OUTCOMES:
Psychometric evaluation of fatigue | 1 day
  The Multidimensional Fatigue Inventory (MFI) is a 20 question self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Each question is graded from 1 ("Yes, that is true") to 5 ("No, that is not true"). Higher scores indicate a higher level of fatigue.
Quality of life impact of fatigue | 1 day
  The functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) evaluates the impact on quality of life of chronic illness.
  This is a questionnaire with 13 questions graded according to a Likert scale ranging from 1 to 5 (1 = quite, 5 = not at all).
Assessment of gait and balance | 1 day
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Assesment of lower limb functional strength | 1 day
  The five-repetition sit-to-stand test (5STS) is a test of lower limb function that measures the fastest time taken to stand five times from a chair with arms folded.
Assesment of walking speed | 1 day
  10 meters gait speed test: measure of the time required to walk 10 meters at the fastest speed possible.
Electromyographic evaluation: temporal recruitment of the motor units. | 1 day
  The evolution of temporal recruitment through the evaluation of the discharge frequency of the motor units.
Electromyographic evaluation: Root Mean Square measurement | 1 day
  The average Root Mean Square (RMS) evolution according to the progress of the fatigability protocol, and its link with the developed force.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgina Piccoli, MD, Principal Investigator — Centre Hospitalier Le Mans, Nephrology Department

IPD SHARING:
Plan to Share IPD: No